CLINICAL TRIAL: NCT00472654
Title: Nutritional Regulation of Bone - Aim 3
Brief Title: The Effect of Vitamin D Supplementation During Caloric Restriction on Intestinal Calcium Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sue A. Shapses, Ph.D., RD, Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG0083; R01AG012161 (NIH); AG012161
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2022-01

CONDITIONS: Weight Loss; Vitamin D or Placebo
Keywords: bone mass; calcium absorption; bone quality; fracture risk
MeSH Terms: conditions — Weight Loss | interventions — Vitamin D; Body Weight Maintenance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- WL (Placebo Comparator)
  Interventions: Behavioral: Weight Loss
- WL + D (Experimental)
  Interventions: Behavioral: Weight Loss; Dietary Supplement: Vitamin D 2500 IU
- WM (Placebo Comparator)
  Interventions: Behavioral: Weight Maintenance
- WM + D (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D 2500 IU; Behavioral: Weight Maintenance

INTERVENTIONS:
Behavioral: Weight Loss — Diet for weight loss for 6 weeks; all weight loss participants will attend 6 weekly counseling sessions (about 50 minutes per session)
  Arms: WL; WL + D
Dietary Supplement: Vitamin D 2500 IU — Daily Vitamin D 2500 IU supplement for 6 weeks
  Arms: WL + D; WM + D
Behavioral: Weight Maintenance — Diet for weight maintenance for 6 weeks
  Arms: WM; WM + D

SUMMARY:
The purpose of this study is to learn how the amount of vitamin D supplementation influences intestinal fractional calcium absorption (a measure of the amount of calcium absorbed).

DETAILED DESCRIPTION:
The extent of change in the amount of calcium that is absorbed with an increase in vitamin D supplementation is not known. This information is important for determining appropriate vitamin D requirements for optimal calcium absorption. During caloric restriction in postmenopausal women, we found that serum parathyroid hormone (PTH) explains 22% of the variance for the reduced calcium absorption (equivalent to 400 IU of Vitamin D per day). It is possible that higher dietary Vitamin D will increase serum 25-hydroxy-Vitamin D (25(OH)D) levels, offset serum PTH and thereby prevent a reduction in calcium absorption. This study seeks to determine if a high Vitamin D intake (a supplement of 2500 IU per day) can increase true fractional calcium absorption (TFCA) in postmenopausal women on a standard high-carbohydrate weight loss diet compared to weight maintenance, with the hypothesis that a high Vitamin D intake will raise serum 25(OH)D and offset the decline in TFCA during caloric restriction (vs. an increase in weight-stable women), and serum PTH will no longer be a major factor explaining changes in TFCA.

Participants will be recruited for both weight loss and weight maintenance, and all will be randomly assigned to take either 2500 IU per day vitamin D supplement or matching placebo. All weight loss participants will attend 5-6 weekly counseling sessions (about 50 minutes per session). All participants will be asked to take a daily vitamin/mineral supplement and, depending on their usual food intake, they may be asked to take a calcium tablet to meet the recommended intake throughout the study period. To measure calcium absorption before and after the 6 weeks of weight loss, participants will go to the study site after an overnight fast where an IV will be placed and the participant will receive an infusion of a stable calcium isotope and consume a 4 oz beverage that also contains a stable isotope of calcium. Blood will be drawn, and then the participant will be asked to collect all urine for the next 24 hours. Body composition (fat, muscle mass, and bone mineral density) will be measured by a dual-energy x-ray absorptiometry (DXA) machine and peripheral quantitative computer tomography (pQCT).

Participants will only be recruited in the winter and spring of each year.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women who are more than 2 years since last menses
* Obese or overweight
* Must live in the geographic vicinity of Rutgers University

Exclusion Criteria:

* Currently on any medication known to influence calcium or bone metabolism, including HRT, or with evidence of diseases known to influence calcium metabolism (i.e. metabolic bone disease, hyperparathyroidism, untreated thyroid disease, significant immune, hepatic, or renal disease, significant cardiac disease [i.e., heart attack or stroke in the past 6 months., abnormal EKG], active malignancy or cancer therapy within the past year)
* History of kidney stones
* Weight gain or weight loss (5% of body wt) within 3 months prior to recruitment
* Participation in other investigational studies during the study period
* Travel for longer than 2 consecutive weeks during the study period
* Usually have a very high or low intake of calcium (more than 1500 or less than 500 mg per day)

Ages: 50 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Changes in Calcium absorption | 6 weeks

SECONDARY OUTCOMES:
Changes in serum and urine bone markers, hormones, glucose, proteins and genes | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sue Shapses, PhD, Principal Investigator — Rutgers University, Nutritional Sciences
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

REFERENCES:
- [Background] Shapses SA, Riedt CS. Bone, body weight, and weight reduction: what are the concerns? J Nutr. 2006 Jun;136(6):1453-6. doi: 10.1093/jn/136.6.1453. PMID 16702302
- [Background] Riedt CS, Cifuentes M, Stahl T, Chowdhury HA, Schlussel Y, Shapses SA. Overweight postmenopausal women lose bone with moderate weight reduction and 1 g/day calcium intake. J Bone Miner Res. 2005 Mar;20(3):455-63. doi: 10.1359/JBMR.041132. Epub 2004 Nov 29. PMID 15746990
- [Background] Cifuentes M, Riedt CS, Brolin RE, Field MP, Sherrell RM, Shapses SA. Weight loss and calcium intake influence calcium absorption in overweight postmenopausal women. Am J Clin Nutr. 2004 Jul;80(1):123-30. doi: 10.1093/ajcn/80.1.123. PMID 15213038
- [Background] Goode LR, Brolin RE, Chowdhury HA, Shapses SA. Bone and gastric bypass surgery: effects of dietary calcium and vitamin D. Obes Res. 2004 Jan;12(1):40-7. doi: 10.1038/oby.2004.7. PMID 14742841
- [Background] Shapses SA, Sukumar D, Schneider SH, Schlussel Y, Brolin RE, Taich L. Hormonal and dietary influences on true fractional calcium absorption in women: role of obesity. Osteoporos Int. 2012 Nov;23(11):2607-14. doi: 10.1007/s00198-012-1901-5. Epub 2012 Jan 27. PMID 22282301
- [Result] Shapses SA, Sukumar D, Schneider SH, Schlussel Y, Sherrell RM, Field MP, Ambia-Sobhan H. Vitamin D supplementation and calcium absorption during caloric restriction: a randomized double-blind trial. Am J Clin Nutr. 2013 Mar;97(3):637-45. doi: 10.3945/ajcn.112.044909. Epub 2013 Jan 30. PMID 23364004